CLINICAL TRIAL: NCT00524329
Title: SYNCHRONISE: Esomeprazole 20 mg Once Daily for Relief of Upper Gastrointestinal Symptoms Associated With Continuous Use of NSAIDs Including COX-2 Selective NSAIDs in Dutch General Practice: The Influence of Risk-Factors for NSAID-Associated GI Damage on Sympton Response
Brief Title: Esomeprazole And Symptomatic Response In Patients With Or Without An Elevated Risk For Non-Steroidal Anti-Inflammatory Drug (NSAID)-Associated GI Damage
Acronym: Synchronise
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind / Medical Science Director, AstraZeneca
Other Study IDs: N13
Record Dates: First submitted 2007-08-29; First posted 2007-09-03 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Heartburn
Keywords: upper GI-symptoms; heartburn; NSAID; risk; PPI; Bloating; Regurgitation
MeSH Terms: conditions — Heartburn; Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to compare the treatment effect in patients with upper gastro-intestinal complaints with an elevated risk for NSAID-associated GI-damage to those without an elevated risk for NSAID-associated damage (as determined by the treating physician).

ELIGIBILITY:
Inclusion Criteria:

* Patient with upper gastro-intestinal complaints (defined as heartburn and/or regurgitation and/or nausea and/or bloated feeling)and treatment with esomeprazole 20mg once daily is started because of this (consult 1). Upper gastro-intestinal complaints are thought to be related to NSAID use
* Patient is using an NSAID** with the following conditions:

  * NSAID use has started at least one week before 1st consultation and is expected to be continued unchanged during the coming period (at least until consult 2)
  * NSAID is taken at least 3 days a week

(**)OTC or Prescription NSAID

(**)Conventional NSAID or COX-2 selective NSAID

Exclusion Criteria:

* Use of a PPI and/or H2RA in the month preceding the study
* A history of reflux disease, not related to NSAID use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at general practitioner
Sampling Method: Non-Probability Sample
Enrollment: 1220 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sellink, Study Director — AstraZeneca; N van den Berk, Study Chair — AstraZeneca